CLINICAL TRIAL: NCT00032903
Title: Oral ST1481 in Adults With Malignant Glioma: a Phase I-II Clinical Trial
Brief Title: This is an Early Study to Investigate the Effect of Gimatecan® in Adults With Malignant Glioma.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sigma-Tau Research, Inc. (Industry)
Collaborators: Rhode Island Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST 01-402
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Malignant Glioma
Keywords: Malignant Glioma, Camptothecin, Pharmacokinetics
MeSH Terms: conditions — Glioma | interventions — ST 1481

INTERVENTIONS:
Drug: Gimatecan® (ST 1481)

SUMMARY:
Gimatecan® is Sigma-Tau Research's new, potent, oral Topoisomerase I inhibitor. Drugs in this class play a crucial role in destroying DNA replication in tumors. We are conducting this study to determine the Maximum Tolerated Dose of our compound. In addition, we plan to assess the drug's ability to affect the evolution of malignant gliomas, when given as a capsule, rather than by intravenous injection.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed diagnosis of a recurrent primary malignant glioma
* Life expectancy of at least 3 months with normal hematological, liver and renal function

Exclusion criteria:

* Pregnant and lactating patients
* Participation in any investigating drug study within 4 weeks preceding treatment start or concurrent treatment with any other anti-cancer therapy
* Gastrointestinal dysfunction that could alter absorption or motility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2002-03; Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States